CLINICAL TRIAL: NCT06401200
Title: Marginal Bone Loss and Soft Tissue Health Around Implants in Selective Laser Melted Versus Milled Cobalt Chromium Bar Retained Mandibular Overdenture:(Randomized Controlled Trial)
Brief Title: Radiographic and Clinical Evaluation In Bar
Acronym: implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Reem Abd El Moatty Abd El Monem, lecturer assistant, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 636; Iman Adel Asfahani (Other: Minia university); Hussein Abd Elhady (Other: Minia UNiversity)
Record Dates: First submitted 2024-04-30; First posted 2024-05-06 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Dental
Keywords: SLM; Milled; Bar overdenture

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1: milled cobalt chromium bar (Active Comparator): 10 completely edentulous patients received two implants at canine region bilaterally (3.7mm diameter- 13mm length), within two weeks after surgery (following early loading protocol), an open tray impression technique was made for bar construction which was designed according to randomization patient enrollment
  Interventions: Other: bar retained implant overdenture
- group 2: Selective laser melted cobalt chromium bar (Experimental): 10 completely edentulous patients received two implants at canine region bilaterally (3.7mm diameter- 13mm length), within two weeks after surgery (following early loading protocol), an open tray impression technique was made for bar construction which was designed according to randomization patient enrollment
  Interventions: Other: bar retained implant overdenture

INTERVENTIONS:
Other: bar retained implant overdenture — use of bar attachment in completely edentulous patient
  Other Names: bar attachment implant mandibular overdenture

SUMMARY:
the aim of this study was to assess the marginal bone loss and soft tissue outcomes of milled and selective laser melted cobalt chromium bar retaining implant mandibular overdenture. Materials and method: twenty completely edentulous patients received new conventional complete dentures. Two implants were placed at mandibular canine areas, patients were randomly allocated into two equal groups: milled co-cr bar group and selective laser melted bar group. Marginal bone loss, modified plaque index (mPI), probing depth (PD) and modified gingival index (mGI) were evaluated at base line, 6 and 12 months follow up visits.

DETAILED DESCRIPTION:
Materials and method: twenty completely edentulous patients received new conventional complete dentures. Two implants were placed at mandibular canine areas, patients were randomly allocated into two equal groups: milled co-cr bar group and selective laser melted bar group. Marginal bone loss, modified plaque index (mPI), probing depth (PD) and modified gingival index (mGI) were evaluated at base line, 6 and 12 months follow up visits.

ELIGIBILITY:
Inclusion Criteria:

* completely edentulous patient.
* age range (50-60) years old.
* adequate bone volume in canine area bilaterally to receive implant of 3.7 mm diameter and 13mm length verified by CBCT for all patients.
* sufficient inter arch space (13-14mm) to accommodate bar construction
* normal maxillo-mandibular relation-ship
* (Angel's class I)
* proper oral hygiene

Exclusion Criteria:

* patients with metabolic or systemic disease that may affect osseointegration.
* history of radiation therapy.
* history of bisphosphonate intake
* heavy smoking and bad habits as bruxism.

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
Radiographic Evaluation (Vertical Marginal bone loss in millimeters) | at 6 and 12 months
  using periapical x-ray with parallel long cone technique from implant shoulder till bony crest

SECONDARY OUTCOMES:
Probing depth in millimeters. | at 0,6 and 12 months
  using sensitive pressure plastic probe in four sites mesial, distal, buccal and lingual
modified Plaque Index. | at 0,6 and 12 months follow up
  using Mombelli charting scale at four aspects (mesial, distal, buccal and lingual)
modified Gingival Index | at base line, 6 and 12 months
  using Apsi charting scale at four sites (mesial, distal, buccal and lingual)

CONTACTS AND LOCATIONS:
Overall Officials: Eman A Asfahani, PHD, Study Chair — Minia University; Hussein A Elhady, PHD, Study Chair — Minia University
Locations (1):
- Minia University, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] El-Asfahani IA, Abd El-Moatty R, Mohamed GF, Hussein HA. Marginal bone loss and soft tissue health around two-implant mandibular overdenture retained with milled versus selective laser melted cobalt chromium bar: a randomized clinical trial. BMC Oral Health. 2024 Oct 4;24(1):1180. doi: 10.1186/s12903-024-04883-6. PMID 39367394